CLINICAL TRIAL: NCT00544700
Title: Bevacizumab Maintenance Versus no Maintenance After Stop of First-line Chemotherapy in Patients With Metastatic Colorectal Cancer. A Randomized Multicenter Phase III Non-inferiority Trial
Brief Title: Bevacizumab in Treating Patients Who Have Undergone First-Line Therapy for Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data collection is completed. As no changes in the endpoints were expected in the future, no further data is needed.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 41/06; SWS-SAKK-41/06; EU-20762; CDR0000569866
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Bevacizumab monotherapy (Active Comparator): Bevacizumab maintenance monotherapy
  Interventions: Biological: bevacizumab
- Arm B: No maintenance (Other): No antitumor treatment until progression
  Interventions: Other: no maintenance

INTERVENTIONS:
Biological: bevacizumab — 7.5 mg/kg i.v. bevacizumab every 21 days until progression or unacceptable toxicity
  Other Names: Avastin®
  Arms: Arm A: Bevacizumab monotherapy
Other: no maintenance — No treatment until progression
  Arms: Arm B: No maintenance

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether giving bevacizumab as maintenance therapy is more effective than observation in treating patients with colorectal cancer.

PURPOSE: This randomized phase III trial is studying bevacizumab to see how well it works in treating patients who have undergone first-line therapy for metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate that time to progression (TTP) without further treatment is not inferior to TTP with maintenance therapy comprising bevacizumab in patients with metastatic colorectal cancer and stable or responding disease after completion of standard first-line chemotherapy/bevacizumab treatment.

Secondary

* To evaluate the safety of bevacizumab maintenance therapy in these patients.
* To assess the long-term cost implications of prolonged treatment with bevacizumab.

OUTLINE: This is a multicenter study. Patients are stratified according to best response during first-line chemotherapy/bevacizumab treatment (complete response and partial response vs stable disease), duration of first-line treatment (16-20 weeks vs 21-24 weeks), type of chemotherapy used during first-line treatment (irinotecan and fluoropyrimidine vs oxaliplatin and fluoropyrimidine vs fluoropyrimidine monotherapy), disease burden (one organ with metastasis vs more than one organ with metastasis), and by participating center.

* Arm I (bevacizumab maintenance therapy): Patients receive bevacizumab IV over 30 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II (no maintenance therapy): Patients receive no further treatment; they are monitored for disease progression.

After completion of study therapy or documentation of disease progression, patients are followed every 3 months for 1 year and then every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic colorectal cancer
* Received prior first-line chemotherapy with oral or intravenous fluoropyrimidine alone or in combination with irinotecan or oxaliplatin

  * Chemotherapy must have been given in combination with a standard dose of bevacizumab for 16-24 weeks as part of first-line treatment for metastatic colorectal cancer
* Stable disease, partial response, or complete response after completion of first-line treatment as documented by abdominal and thoracic CT scan, MRI, or x-ray within the past 21 days
* No clinical symptoms or history of CNS metastases

  * No imaging required in asymptomatic patients

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Serum creatinine < 2.0 mg/dL or 177 μmol/L
* Proteinuria < 2+ by urine dipstick OR urine protein ≤ 1 g by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* Must have basic health insurance with a Swiss health insurance company
* Patients must be compliant and in geographic proximity to allow proper staging and follow-up
* No medical reason that prohibits further bevacizumab treatment, including any of the following:

  * Uncontrolled hypertension (systolic blood pressure [BP] > 150 mm Hg and/or diastolic BP > 100 mm Hg) or clinically significant (i.e., active) cardiovascular disease
  * Serious non-healing wound, active peptic ulcer, or non-healing bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
  * History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
* No serious underlying medical condition that, in the judgment of the investigator, could further impair the ability of the patient to participate in the trial (e.g., active autoimmune disease or uncontrolled diabetes)
* No psychiatric disorder that would preclude patient understanding of study-related topics or giving informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior bevacizumab
* No prior anti-EGFR treatment (e.g., cetuximab) during first-line therapy
* No anticipation of concurrent major surgery (e.g., resection) or ablation of metastases
* No concurrent elective major surgery
* No concurrent daily aspirin exceeding 325 mg/day or clopidogrel exceeding 75 mg/day

  * Lower doses of the drugs noted above, or non-steroidal anti-inflammatory drugs with activity on platelets and gastric mucosa, or dipyridamole are allowed if given at a stable dose for ≥ 2 weeks prior to study entry
* No other concurrent experimental drugs or anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2007-11-26 (Actual); Primary Completion 2013-01-21 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | From randomization until documented progressive disease or death due to tumor.
  TTP will be calculated from randomization until documented PD or death due to tumor.

SECONDARY OUTCOMES:
Overall survival (OS) | OS will be calculated from start of first-line treatment until death. Additionally, OS will be calculated from randomization until death.
  OS will be calculated from start of first-line treatment until death. Additionally, OS will be calculated from randomization until death.
Progression-free survival (PFS) | From start of first-line treatment until documented PD or death, whichever occurs first.
  PFS will be calculated from start of first-line treatment until documented PD or death, whichever occurs first. Additionally, PFS will be calculated from randomization until documented PD or death, whichever occurs first.
Adverse events (AE) | Predefined AEs and AEs ≥ grade 3 will be assessed according to NCI CTCAE v3.0.
  Predefined AEs and AEs ≥ grade 3 will be assessed according to NCI CTCAE v3.0.
Long-term bevacizumab treatment costs | Estimated for the time period between randomization and the end of the follow-up phase (lasting maximal 5 years).
  Costs of bevacizumab treatment, including additional treatments and/or hospitalisations related to bevacizumab, as well as other anticancer treatments and their related hospitalisations, will be estimated for the time period between randomization and the end of the follow-up phase (lasting maximal 5 years) from information collected on the CRFs during trial treatment and follow-up phase.

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koeberle, MD, Study Chair — St. Claraspital Basel; Peter Moosmann, MD, Study Chair — Kantonsspital Aarau
Locations (29):
- Switzerland (29):
  - Kantonsspital Aarau, Aarau
  - Hirslanden Klinik Aarau, Aarau
  - Kantonsspital Baden, Baden
  - St. Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - Spital Buelach, Bülach
  - AndreasKlinik Cham Zug, Cham
  - Kantonsspital Graubuenden, Chur
  - Hopital Fribourgeois, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Kantonsspital Luzern, Luzerne
  - Onkologie Zentrum am Spital Maennedorf, Männedorf
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopital Regional de Sion-Herens-Conthey, Sion
  - Regionalspital, Thun
  - Spital Uster, Uster
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum Klinik im Park, Zurich
  - Klinik Hirslanden, Zurich
  - Stadtspital Waid, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koeberle D, Betticher DC, von Moos R, Dietrich D, Brauchli P, Baertschi D, Matter K, Winterhalder R, Borner M, Anchisi S, Moosmann P, Kollar A, Saletti P, Roth A, Frueh M, Kueng M, Popescu RA, Schacher S, Hess V, Herrmann R. Bevacizumab continuation versus no continuation after first-line chemotherapy plus bevacizumab in patients with metastatic colorectal cancer: a randomized phase III non-inferiority trial (SAKK 41/06). Ann Oncol. 2015 Apr;26(4):709-714. doi: 10.1093/annonc/mdv011. Epub 2015 Jan 20. PMID 25605741